CLINICAL TRIAL: NCT01048450
Title: A Multi-Center Retrospective Review of Resectional Arthroplasty, Arthrodesis and, Hemi-Metallic Joint Implants in the Surgical Treatment of End Stage Hallux Rigidus
Brief Title: Surgical Treatment for Hallux Rigidus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Foot and Ankle Surgeons (Other)
Responsible Party: Paul J Kim, DPM, FACFAS, Associate Professor, American College of Foot and Ankle Surgeons
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0709-1
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2010-01

CONDITIONS: Hallux Limitus; Hallux Rigidus
Keywords: arthritis; degeneration
MeSH Terms: conditions — Hallux Limitus; Hallux Rigidus; Arthritis | interventions — Arthrodesis; Joint Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Those who were diagnosed with hallux limitus/rigidus (end stage degeneration at the 1st metatarsal phalangeal joint)
  Interventions: Radiation: Joint Resection- Keller Procedure; Procedure: Joint Fusion; Procedure: Hemi-metallic Joint Implant

INTERVENTIONS:
Radiation: Joint Resection- Keller Procedure — These subjects had received a surgical intervention of removing the proximal portion of the proximal phalanx of the hallux
  Other Names: Keller Arthoplasty
Procedure: Joint Fusion — Those who had a surgical intervention of fusion of the 1st metatarsal phalangeal joint.
  Other Names: Arthrodesis
Procedure: Hemi-metallic Joint Implant — Those who had a surgical procedure of a hemi-metallic joint implant
  Other Names: Joint Implant

SUMMARY:
The purpose of this study is to examine the long-term outcomes for the surgical treatment of end stage degeneration in the big toe joint.

DETAILED DESCRIPTION:
Hallux rigidus is a degenerative process that occurs in the first metatarsophalangeal joint (MTPJ). There are a variety of surgical treatment options available for its treatment including joint sparing and joint destructive procedures. Patients with end stage arthritis are often given several surgical options for the treatment of the first MTPJ. The procedures are correlated to the patient's age, type of shoe gear, activity level, Body Mass Index, degree of arthritis, desire for joint mobility and bone density. This proposal outlines a retrospective study on the long-term efficacy of joint resection, joint fusion, and hemi-metallic first MTPJ implants. A multi-center study of 300 subjects who received surgical repair for end stage arthritis of the first MTPJ will be evaluated. Subjective assessment for pain, function and alignment as well as objective radiographic evaluation will be performed. Further, the frequency and types of adverse events associated with the three surgical techniques will be assessed. The results of this study will provide valuable information to foot and ankle surgeons in making appropriate decisions regarding the treatment options for end stage hallux rigidus.

ELIGIBILITY:
Inclusion Criteria:

* End stage hallux limitus/rigidus
* Status post 1 year since having the surgery
* Must have had a joint resection, fusion, or hemi-metallic implant

Exclusion Criteria:

* History of seropositive or seronegative arthritis
* Have had a primary surgery before then had one of the above surgeries performed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Subjective: pain, function, alignment | At least 1 year after surgical intervention

SECONDARY OUTCOMES:
Frequency and types of undesired effects | At least 1 year after surgical intervention
Demographic data and trends | At least 1 year after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Kim, DPM, Study Director — American College of Foot & Ankle Surgeons
Locations (6):
- United States (6):
  - Foot & Ankle Center of Northern Colorado, Greeley, Colorado
  - Capitol Orthopaedics & SPorts Medicine, Des Moines, Iowa
  - Scituate Podiatry Group, Scituate, Massachusetts
  - Michigan Foot & Ankle Center, Southfield, Michigan
  - Ankle and Foot Care Centers, Youngstown, Ohio
  - Marc Kravettte, Seattle, Washington

REFERENCES:
- [Background] Gibson JN, Thomson CE. Arthrodesis or total replacement arthroplasty for hallux rigidus: a randomized controlled trial. Foot Ankle Int. 2005 Sep;26(9):680-90. doi: 10.1177/107110070502600904. PMID 16174497
- [Background] Raikin SM, Ahmad J. Comparison of arthrodesis and metallic hemiarthroplasty of the hallux metatarsophalangeal joint. Surgical technique. J Bone Joint Surg Am. 2008 Oct;90 Suppl 2 Pt 2:171-80. doi: 10.2106/JBJS.H.00368. PMID 18829931
- See also: Sponsor's Web site — http://www.acfas.org